CLINICAL TRIAL: NCT07200466
Title: ENDORISK Clinical Implementation Study
Brief Title: Individualised Endometrial Cancer Risk Stratification by Bayesian Prediction Model (ENDORISK), Optimizing Clinical Implementation
Acronym: ENDORISK-I
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Elisabeth-TweeSteden Ziekenhuis (Other); Amphia Hospital (Other); Catharina Ziekenhuis Eindhoven (Other); Elkerliek Hospital (Other); St. Anna Ziekenhuis, Geldrop, Netherlands (Other); Jeroen Bosch Ziekenhuis, s'-Hertogenbosch (Unknown); Rijnstate Hospital (Other); Canisius Wilhelmina Ziekenhuis (CWZ) (Unknown); Maxima Medical Center (Other); Bernhoven Hospital (Other); Maas Hospital Pantein (Other); Slingeland Hospital (Other); Streekziekenhuis Koningin Beatrix (Unknown); Gelderse Vallei Hospital (Other); Comprehensive Cancer Centre The Netherlands (Other); Stichting PAMM (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL86300.000.24; 14032 (Other Grant/Funding Number: Koningin Wilhelmina Fonds voor Nederlandse Kankerbestrijding)
Record Dates: First submitted 2025-07-23; First posted 2025-10-01 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-07

CONDITIONS: Endometrial Cancer
Keywords: ENDORISK; Endometrial Cancer; surgical staging; risk stratification; lymph node metastases; lymphadenectomy; sentinel node
MeSH Terms: conditions — Endometrial Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Intervention Model Description: Patients will receive a personalized treatment plan based on the risk of lymph node metastases as predicted by the ENDORISK model. Patients with low grade endometrial cancer (EC) (grade I-II) at high risk of lymph node metastases might therefore undergo additional surgical staging, through either sentinel lymph node procedure or lymphadenectomy. Patients with low grade EC (grade I-II) at low-risk of lymph node metastases are counselled to undergo standard treatment, which involves hysterectomy with bilateral salpingo-oophorectomy. Patients with high grade EC (grade III), receive their personalized risk but will undergo standard care to further validate the ENDORISK model in this group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The control arm is a group of patients from our previous 'evaluation of care' study which underwent standard care for endometrial cancer between march of 2022 and the start of the ENDORISK-I study. This group serves as a control group for the intervention arm.
- Intervention (Experimental): The intervention group are patients receiving a personalized risk on lymph node metastases as predicted by the ENDORISK model, they also receive a treatment plan (hysterectomy + bilateral salpingo-oophorectomy with or without lymph node surgery) based on this personalized risk.
  Interventions: Diagnostic Test: ENDORISK personalized risk assesment for lymph node metastases in endometrial cancer.

INTERVENTIONS:
Diagnostic Test: ENDORISK personalized risk assesment for lymph node metastases in endometrial cancer. — The intervention group are patients receiving a personalized risk on lymph node metastases as predicted by the ENDORISK model, they also receive a treatment plan (hysterectomy + bilateral salpingo-oophorectomy with or without lymph node surgery) based on this personalized risk.
  Arms: Intervention

SUMMARY:
Rationale: Preoperative identification of patients at risk for lymph node metastasis (LNM) is challenging in endometrial cancer (EC). Therefore, a Bayesian network model called ENDORISK was developed and validated in three external cohorts to improve preoperative risk stratification. The next step is to implement and evaluate whether use of the model improves daily clinical practice. Objective: The ENDORISK implementation (ENDORISK-I) study aims to prospectively evaluate whether implementation of ENDORISK in daily clinical practice improves preoperative risk stratification. Study design: A stepped wedge non inferiority study in which two oncology regions will consecutively start implementation of ENDORISK with one year interval. The ENDORISK model will be filled in and used in preoperative treatment counselling. Results will be compared to current standard clinical care which is prospectively evaluated in both regions since March 2022 in the 'evaluation of care in endometrial cancer' study (2021-7400). Study population: all consecutive patients recently diagnosed with early stage EC who are eligible for surgical treatment, who understand Dutch and are able to fill in a digital or paper questionnaire can be included. Main study parameters/endpoints: The ENDORISK implementation (ENDORISK-I) study aims to prospectively evaluate implementation of ENDORISK in daily clinical practice by investigating:

* The proportion of identified LNM in patients with lymph node staging (positive predictive value (PPV)) compared to standard care
* Proportion of patients who decide to have lymph node status assessed in ENDORISK care compared to standard care
* Preoperative information provision for patients and shared-decision making with the use of ENDORISK compared to standard care
* Patients' disease- specific-, overall survival, and health-related quality of life compared to standard care
* Patients' and doctors' use of and experiences with the ENDORISK-model
* Impact of ENDORISK on regional care costs

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with early stage (FIGO stage I-II) endometrial carcinoma (every grade permitted)
* Eligible for primary surgical treatment (neo-adjuvant therapy is permitted)

Exclusion Criteria:

* Unable to give informed consent
* No understanding of Dutch or English language
* Rare types of endometrial cancer, such as endometrial stroma cell sarcoma

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 735 (Estimated)
Dates: Start 2025-10-23 (Actual); Primary Completion 2027-10-16 (Estimated); Study Completion 2032-10-16 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who decide to have lymph node status assessed in ENDORISK care compared to standard care. | from enrolment to surgery
Proportion of patients with lymph node metastases within patients undergoing lymph node staging (the positive predictive value) in ENDORISK care | From enrolment to time of surgery
  The lymph node metastases in patients undergoing lymph node staging will be determined by pathology report on the surgical specimen. The positive predicting value will be compared to the positive predictive value of standard care.
Preoperative information provision for patients and shared-decision making with the use of ENDORISK compared to standard care, measured by questionnaires. | From enrolment to 12 weeks post-operatively
  Information provision score: Questionnaire EORTC Quality of Life Questionnaire (QLQ)-INFO25 with additional questions specific to ENDORISK use.
  Shared-decision making score: Shared Decision Making Questionnaire SDM-Q-9 with additional questions specific to ENDORISK use

SECONDARY OUTCOMES:
Patients' 5-year disease- specific-, overall survival (DSS, OS), compared to standard care; | from enrolment to 5-year post surgery
Health related quality of life (HRQoL) compared to standard care | 12 weeks after primary surgery
  as measured by questionnaire: EORTC Quality of life questionnaire (QLQ) -C30
Health-related quality of life (HRQoL) compared to standard care | 12 months after primary surgery
  as measured by questionnaire: EORTC QLQ-C30
Treatment-related morbidity compared to standard care | 12 weeks after primary surgery
  As measured by questionnaire: EORTC QLQ- Endometrial cancer (EN) 24
Treatment related morbidity compared to standard care | 12 months after primary surgery
  As measured by questionnaire: EORTC QLQ-EN24 and questionnaires about lymphoedema: EORTC IL76 & Lymphoedema quality of Life (LYMQOL)
Clinicians' experiences with ENDORISK care | at baseline
  Questionnaire at baseline
Clinicians' experiences with ENDORISK care | 9 months after start of inclusions
  Questionnaire at 9 months
Clinicians' experiences with ENDORISK care | 18 months after start of inclusions
  Questionnaire at 18 months
Clinicians' experiences with ENDORISK care | Within 1 year of start of the inclusion period in their hospital.
  In depth interviews with a sample of participating clinicians to evaluate user experiences.
Impact of ENDORISK on regional care costs | from enrolment to the end of inclusions

OTHER OUTCOMES:
Charlson-index | 12 weeks after primary surgery
  Charlson-index as reported by participants and as reported by clinician/researcher from patient records
Health literacy | 12 weeks after primary surgery
  Health Literacy as reported by participants through a questionnaire

CONTACTS AND LOCATIONS:
Locations (14):
- Netherlands (14):
  - Rijnstate, Arnhem, Gelderland
  - Slingeland Hospital, Doetinchem, Gelderland
  - Gelderse Vallei, Ede, Gelderland
  - Radboudumc, Nijmegen, Gelderland
  - Canisius Wilhelmina Ziekenhuis (CWZ), Nijmegen, Gelderland
  - Streekziekenhuis Koningin Beatrix, Winterswijk, Gelderland
  - Jeroen Bosch Hospital, 's-Hertogenbosch, North Brabant
  - Amphia, Breda, North Brabant
  - Catharina Hospital, Eindhoven, North Brabant
  - St. Anna Hospital, Geldrop, North Brabant
  - Elkerliek Hospital, Helmond, North Brabant
  - Elisabeth-Tweesteden Hospital, Tilburg, North Brabant
  - Bernhoven Hospital, Uden, North Brabant
  - Maxima Medical Center, Veldhoven, North Brabant

IPD SHARING:
Plan to Share IPD: Yes
Only anonymized datasets (without patient numbers, date of birth or name) will be shared with other people relevant to the study or relevant to additional studies as reported in the patient information folder.
  Patients are requested whether or not they give permission to use anonymized data from this study for further research into cervical cancer.
Supporting Information: Study Protocol
Time Frame: IPD will be available after the end of the study.
Access Criteria: Researchers within the RadboudUMC will be able to get access upon request and review of research aim/protocol

REFERENCES:
- [Background] Vinklerova P, Ovesna P, Hausnerova J, Pijnenborg JMA, Lucas PJF, Reijnen C, Vrede S, Weinberger V. External validation study of endometrial cancer preoperative risk stratification model (ENDORISK). Front Oncol. 2022 Aug 3;12:939226. doi: 10.3389/fonc.2022.939226. eCollection 2022. PMID 35992828
- [Background] Reijnen C, Gogou E, Visser NCM, Engerud H, Ramjith J, van der Putten LJM, van de Vijver K, Santacana M, Bronsert P, Bulten J, Hirschfeld M, Colas E, Gil-Moreno A, Reques A, Mancebo G, Krakstad C, Trovik J, Haldorsen IS, Huvila J, Koskas M, Weinberger V, Bednarikova M, Hausnerova J, van der Wurff AAM, Matias-Guiu X, Amant F; ENITEC Consortium; Massuger LFAG, Snijders MPLM, Kusters-Vandevelde HVN, Lucas PJF, Pijnenborg JMA. Preoperative risk stratification in endometrial cancer (ENDORISK) by a Bayesian network model: A development and validation study. PLoS Med. 2020 May 15;17(5):e1003111. doi: 10.1371/journal.pmed.1003111. eCollection 2020 May. PMID 32413043
- [Background] Grube M, Reijnen C, Lucas PJF, Kommoss F, Kommoss FKF, Brucker SY, Walter CB, Oberlechner E, Kramer B, Andress J, Neis F, Staebler A, Pijnenborg JMA, Kommoss S. Improved preoperative risk stratification in endometrial carcinoma patients: external validation of the ENDORISK Bayesian network model in a large population-based case series. J Cancer Res Clin Oncol. 2023 Jul;149(7):3361-3369. doi: 10.1007/s00432-022-04218-4. Epub 2022 Aug 8. PMID 35939115
- See also: ENDORISK website with information relating to the ENDORISK model and the research team — https://www.endorisk.eu/

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-08-26): https://cdn.clinicaltrials.gov/large-docs/66/NCT07200466/Prot_SAP_000.pdf
  • Informed Consent Form (2025-08-26): https://cdn.clinicaltrials.gov/large-docs/66/NCT07200466/ICF_001.pdf